CLINICAL TRIAL: NCT06229132
Title: Building Mobile HIV Prevention and Mental Health Support in Low-resource Settings
Brief Title: Mental Health Support for Transgender and Gender-expansive Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Yale University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Corina Lelutiu-Weinberger, Associate Professor of Health Sciences Research, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAU2518-TGD; R01MH116829 (NIH)
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Results first posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Transgender; Depression; Anxiety; Suicidality; HIV
Keywords: Transgender; Gender diverse; Mental health
MeSH Terms: conditions — Depression; Anxiety Disorders; Suicidal Ideation; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LGBTQ-affirmative CBT treatment (Other): LGBTQ-affirmative CBT includes client case conceptualizations to personalize treatment delivery and functional relevance. Modules raise awareness of the impact of sexual minority stress on mental, behavioral, and sexual health; instill cognitive flexibility toward minority stress cognitions; and reduce maladaptive avoidance tendencies rooted in minority stress. The treatment is guided by six principles: (1) normalizing mood and anxiety as a common response to LGBTQ-related stress; (2) challenging persistent, inflexible LGBTQ-related stress-induced cognitions; (3) encouraging assertive behavior and open self-expression in safe situations to effectively cope with the consequences of LGBTQ-related stress; (4) validating LGBTQ clients' unique strengths; (5) building authentic relationships as an essential resource for LGBTQ people's mental health; and (6) recognizing intersectional identities as a source of stress and resilience. The intervention consists of 16 sessions delivered on Zoom.
  Interventions: Behavioral: LGBTQ-affirmative CBT for transgender individuals

INTERVENTIONS:
Behavioral: LGBTQ-affirmative CBT for transgender individuals — The intervention addresses unique stressors encountered by transgender individuals due to discrimination and lack of adequate and affirming healthcare resources.

SUMMARY:
This study will evaluate an intervention's feasibility, acceptability and efficacy potential in a one-arm trial with Romanian transgender and gender diverse (e.g., gender non-binary) (TGD) individuals who report depression or anxiety. The intervention will consist of 16 1-hour sessions delivered by our trained therapists on Zoom. These sessions are based on 6 principles of LGBTQ-affirming CBT, as follows: (1) normalizing mood and anxiety as a common response to LGBTQ related stress; (2) challenging persistent, inflexible LGBQ-related stress-induced cognitions; (3) encouraging assertive behavior and open self-expression to effectively cope with the consequences of LGBTQ-related stress; (4) validating lesbian, gay, bisexual, and transgender (LGBTQ) clients' unique strengths; (5) building authentic relationships as an essential resource for LGBTQ people's mental health; and (6) recognizing intersectional identities as a source of stress and resilience.

DETAILED DESCRIPTION:
Transgender and gender diverse (e.g., gender non-binary) (TGD) individuals remain a hidden group in the Central Eastern European (CEE) country of Romania, with few protections, few equal rights, and many unmet needs. Emerging research with TGD persons in the region indicates that TGD Romanians report particularly high rates of HIV, depression, and hazardous alcohol use, primarily driven by the country's high structural stigma. Romania's healthcare system has little expertise for addressing these syndemic health threats. No targeted needs assessments or interventions exist to date in order to remedy these adversities and promote the wellbeing of TGD in Romania, or anywhere in CEE - the region with the fastest-growing HIV epidemic in the world. In response, the investigators propose to create and pilot-test the first intervention in CEE to address the sexual, mental, and behavioral health of TGD people. In Aim 1, the investigators will identify unique needs of TGD Romanians via interviews. Findings will be used in Aim 2 to modify an intervention manual to address gender minority stress and other TGD-specific determinants of mental health, hazardous alcohol use, and HIV risk. The intervention will be based on a Romanian-adapted EQuIP (Empowering Queer Identities in Psychotherapy) intervention d developed and successfully tested by our team in several global regions (e.g., the U.S., China). In Aim 3, the investigators will evaluate the adapted intervention's feasibility, acceptability, and efficacy potential in a one-arm trial with 25 TGD Romanians. By extending the intervention research to at-risk TGD populations, the investigators will ensure more equitable access to the interventions and embed them within a national infrastructure increasingly eager for and capable of reaching the full diversity of the Romanian LGBTQ population to address its currently unmet needs.

ELIGIBILITY:
Inclusion Criteria:

1. report an identity as transgender or gender expansive (e.g., gender non-binary) and a gender that is different from their assigned sex at birth;
2. be ≥18 years old;
3. report a score of ≥2.5 on either the two items measuring depression symptoms or the two items measuring anxiety symptoms using the Brief Symptom Inventory (BSI-4); and
4. reside in Romania for the duration of the study (approximately 6 months).

Exclusion Criteria:

1. active suicidality, mania, or psychosis and
2. having received CBT in the prior 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Individuals who report an identity as transgender or gender expansive (e.g., gender non-binary) and a gender that is different from their assigned sex at birth will be included.
Enrollment: 25 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corina Lelutiu-Weinberger, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University School of Nursing, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- TGE Individuals: Transgender and gender expansive (TGE) individuals living in Romania
Period: Overall Study
Arm/Group | TGE Individuals
Started | 25
Completed | 22
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | TGE Individuals
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.16 (6.39)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Sex assigned at birth
  Participants
    Female | 13
    Male | 10
    Intersex | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Romanian | 21
  Roma | 1
  Other | 3
Region of Enrollment [Number; unit: participants]
  Romania | 25
Gender identity [Count of Participants; unit: Participants]
  Transgender woman | 11
  Transgender man | 10
  Nonbinary (e.g., genderqueer, agender, gender fluid) | 4
Sexual orientation [Count of Participants; unit: Participants]
  Bisexual | 5
  Demisexual | 1
  Gay | 1
  Heterosexual | 8
  Pansexual | 4
  Queer | 6
Educational attainment [Count of Participants; unit: Participants]
  High school or less | 12
  Some college | 4
  College degree | 7
  Graduate degree | 2

OUTCOME MEASURES:

1. Primary Outcome: Depression: Score on the Overall Depression Severity & Impairment Scale (ODSIS)
Description: Participants will complete the Overall Depression Severity & Impairment Scale (ODSIS) to assess past-week frequency, severity, and impairment related to depression symptoms. The ODSIS is comprised of five items (e.g., "In the past week, how often have you felt depressed?") each measured on a five-point scale ranging from 0 (no depression in the past week) to 4 (constant depression: felt depressed all of the time). Item scores will be summed to obtain a total score ranging from 0 (min) to 20 (max), with a higher total score indicating greater depressive symptoms (worse outcome).
Time Frame: Measured at baseline and 5 months post-baseline
Population: 25 participants completed baseline measures, and 22 participants completed the 5-month follow up. Data for this outcome measure was not collected from those 3 participants who did not complete the 5-month follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TGE Individuals
Number analyzed (Participants) | 25
score on a scale
  Baseline | 9.68 (4.96)
  5 months post-baseline: number analyzed (Participants) | 22
  5 months post-baseline | 4.82 (5.04)

2. Secondary Outcome: Anxiety: Score on the Overall Anxiety Severity & Impairment Scale (OASIS)
Description: Participants will complete the Overall Anxiety Severity & Impairment Scale (OASIS), which is comprised of five items (e.g., "In the past week, how often have you felt anxious?") measured on a five-point scale ranging from 0 (no anxiety in the past week) to 4 (constant anxiety: felt anxious all of the time and never really relaxed). Item scores will be summed to obtain a total score ranging from 0 (min) to 20 (max), with a higher total score indicating greater anxiety symptoms (worse outcome).
Time Frame: Measured at baseline and 5 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TGE Individuals
Number analyzed (Participants) | 25
score on a scale
  Baseline | 10.1 (3.72)
  5 months post-baseline: number analyzed (Participants) | 22
  5 months post-baseline | 5.05 (4.69)

3. Secondary Outcome: Psychological Distress: Score on the Brief Symptom Inventory (BSI)
Description: Psychological distress will be assessed using the Brief Symptom Inventory (BSI) consisting of 18 items scored from 0 (not at all) to 4 (extremely) regarding the extent to which depression symptoms (e.g., "feeling hopeless about the future"), anxiety symptoms (e.g., "feeling tense or keyed up"), and somatization symptoms (e.g., "feeling weak in parts of your body") have distressed the respondent over the past week. Item scores will be averaged to obtain a total score ranging from 0 (min) to 4 (max), with a higher total score indicating greater psychological distress (worse outcome).
Time Frame: Measured at baseline and 5 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TGE Individuals
Number analyzed (Participants) | 25
score on a scale
  Baseline | 1.46 (0.729)
  5 months post-baseline: number analyzed (Participants) | 22
  5 months post-baseline | 1.11 (0.745)

4. Secondary Outcome: Suicidal Ideation: Score on the Suicidal Ideation Attributes Scale (SIDAS)
Description: The Suicidal Ideation Attributes Scale (SIDAS) will assess participants' past-month suicidal thoughts and severity on a ten-point scale ranging from 0 (never or not at all) to 10 (always or extremely). Participants who report no ideation (score of 0) in response to the first item ("In the past month, how often have you had thoughts about suicide") are not presented with subsequent four items regarding the severity of these thoughts and their total score will be recoded as 0. Total scores are calculated as the sum of the five items, with the controllability item reverse scored (i.e., original score of 10 reverse scored as 0, original score of 9 reverse scored as 1, …, original score of 0 reverse scored as 10). Total scores range from 0 (min) to 50 (max), with a higher total score indicating greater suicidal ideation (worse outcome).
Time Frame: Measured at baseline and 5 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TGE Individuals
Number analyzed (Participants) | 25
score on a scale
  Baseline | 8.00 (10.70)
  5 months post-baseline: number analyzed (Participants) | 22
  5 months post-baseline | 4.50 (7.97)

5. Secondary Outcome: Hazardous Drinking: Score on the Alcohol Use Disorders Identification Test (AUDIT-C)
Description: The three-item Alcohol Use Disorders Identification Test (AUDIT-C) will capture frequency of drinking over the past year (e.g., "How often during the past year did you have a drink containing alcohol?"), with response options between 0 (never) and 4 (four or more times per week). Item scores are summed to obtain a total score ranging from 0 (min) to 12 (max), where scores of 0 reflect no alcohol use. The higher the total score, the more likely it is that the respondent's drinking is affecting his/her health and safety (a worse outcome).
Time Frame: Measured at baseline and 5 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TGE Individuals
Number analyzed (Participants) | 25
score on a scale
  Baseline | 2.92 (2.25)
  5 months post-baseline: number analyzed (Participants) | 22
  5 months post-baseline | 2.18 (1.97)

6. Secondary Outcome: Anticipated Stigma: Score on the Negative Expectations for Future Events Subscale of the Gender Minority Stress and Resilience Measure (GMSR)
Description: Responses to each item on the 9-item Negative Expectations for Future Events subscale of the Gender Minority Stress and Resilience Measure (GMSR) are scored on a five-point scale from 0 (strongly disagree) to 4 (strongly agree). An example item includes: "If I express my gender history, employers would not hire me." The items will be summed to obtain a total score ranging from 0 (min) to 36 (max), with a higher total score indicating greater fear of future rejection based on gender identity (worse outcome).
Time Frame: Measured at baseline and 5 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TGE Individuals
Number analyzed (Participants) | 25
score on a scale
  Baseline | 25.7 (5.73)
  5 months post-baseline: number analyzed (Participants) | 22
  5 months post-baseline | 19.9 (8.80)

7. Secondary Outcome: Internalized Stigma: Score on the Internalized Transphobia Subscale of the Gender Minority Stress and Resilience Measure (GMSR)
Description: The eight items of the Internalized Transphobia subscale of the Gender Minority Stress and Resilience Measure (GMSR) are each scored on a five-point scale from 0 (strongly disagree) to 4 (strongly agree). An example item includes: "I resent my gender identity or expression." Item scores will be summed to produce a total score ranging from 0 (min) to 32 (max), where a higher total score indicates greater internalized transphobia (worse outcome).
Time Frame: Measured at baseline and 5 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TGE Individuals
Number analyzed (Participants) | 25
score on a scale
  Baseline | 14.0 (9.40)
  5 months post-baseline: number analyzed (Participants) | 22
  5 months post-baseline | 12.3 (9.25)

8. Secondary Outcome: Gender Identity Rumination: Score on the Gender Identity Reflection and Rumination Scale (GRRS)
Description: The 15-item Gender Identity Reflection and Rumination Scale (GRRS) assesses the extent to which respondents think about their gender identity in various ways. Responses to items are scored on a four-point scale from 1 (almost never) to 4 (almost always). An example item is: "Analyze how my experience of my gender identity shapes who I am." Item scores are summed to obtain an overall score ranging from 15 to 60, where a higher total score indicates more rumination (worse outcome).
Time Frame: Measured at baseline and 5 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TGE Individuals
Number analyzed (Participants) | 25
score on a scale
  Baseline | 38.1 (10.1)
  5 months post-baseline: number analyzed (Participants) | 22
  5 months post-baseline | 34.5 (7.59)

9. Secondary Outcome: Pride: Score on the Pride Subscale of the Gender Minority Stress and Resilience Measure (GMSR)
Description: Responses to the eight items that make up the Pride subscale of the Gender Minority Stress and Resilience Measure (GMSR) are scored on a five-point scale from 0 (strongly disagree) to 4 (strongly agree). An example item is: "My gender identity or expression makes me feel special and unique." Item scores will be summed to produce an overall score ranging from 0 (min) to 32 (max), where a higher overall score indicate greater pride in one's gender identity (better outcome).
Time Frame: Measured at baseline and 5 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TGE Individuals
Number analyzed (Participants) | 25
score on a scale
  Baseline | 14.7 (6.69)
  5 months post-baseline: number analyzed (Participants) | 22
  5 months post-baseline | 14.6 (8.16)

10. Secondary Outcome: Community Connectedness: Score on the Community Connectedness Subscale of the Gender Minority Stress and Resilience Measure (GMSR)
Description: Responses to items on the five-item Community Connectedness subscale of the Gender Minority Stress and Resilience Measure (GMSR) are scored on a five-point scale from 0 (strongly disagree) to 4 (strongly agree). An example item is: "I feel part of a community of people who share my gender identity." Item scores will be summed to produce a an overall score ranging from 0 (min) to 20 (max), where a higher overall score indicates greater connectedness with people who share one's gender identity (better outcome).
Time Frame: Measured at baseline and 5 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TGE Individuals
Number analyzed (Participants) | 25
score on a scale
  Baseline | 12.2 (4.78)
  5 months post-baseline: number analyzed (Participants) | 22
  5 months post-baseline | 12.7 (4.41)

11. Secondary Outcome: Emotion Dysregulation: Score on the Difficulties in Emotion Regulation Scale-Short Form (DERS-SF)
Description: The 18-item Difficulties in Emotion Regulation Scale-Short Form (DERS-SF) assessed frequency of emotion dysregulation on a five-point scale from 1 (almost never) to 5 (almost always). An example item is: "When I'm upset, I acknowledge my emotions." Item scores are averaged to produce an overall score ranging from 1 (min) to 5 (max), where a higher overall score indicates greater difficulties regulating emotions (worse outcome).
Time Frame: Measured at baseline and 5 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TGE Individuals
Number analyzed (Participants) | 25
score on a scale
  Baseline | 2.90 (0.60)
  5 months post-baseline: number analyzed (Participants) | 22
  5 months post-baseline | 2.61 (0.73)

12. Secondary Outcome: Social Support: Score on the Multidimensional Scale of Perceived Social Support (MSPSS)
Description: The 12-item Multidimensional Scale of Perceived Social Support (MSPSS) assesses perceived support from family, friends, and significant others on an seven-point scale from 1 (very strongly disagree) to 7 (very strongly agree). An example item is: "There is a special person who is around when I am need." Item scores are averaged to obtain an overall score ranging from 1 (min) to 7 (max), where a higher overall score indicate greater social support (better outcome).
Time Frame: Measured at baseline and 5 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TGE Individuals
Number analyzed (Participants) | 25
score on a scale
  Baseline | 4.40 (1.03)
  5 months post-baseline: number analyzed (Participants) | 22
  5 months post-baseline | 4.82 (1.23)

13. Secondary Outcome: Unassertiveness: Score on the Simple Rathus Assertiveness Schedule-Short Form (SRAS-SF)
Description: The 19-item Simple Rathus Assertiveness Schedule-Short Form (SRAS-SF) assesses respondents' assertive and unassertive behavior on a six-point scale from 1 (very uncharacteristic of me) to 6 (very characteristic of me) with certain items reverse scored. An example item is: "I strive to get ahead as much as other people in my position." Item scores will be summed to obtain a total score from 19 (min) to 114 (max), where a higher total score indicates greater unassertive behavior (worse outcome).
Time Frame: Measured at baseline and 5 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TGE Individuals
Number analyzed (Participants) | 25
score on a scale
  Baseline | 72.0 (11.1)
  5 months post-baseline: number analyzed (Participants) | 22
  5 months post-baseline | 67.3 (9.45)

14. Secondary Outcome: Rumination: Score on the Brooding Subscale From the Ruminative Responses Scale (RRS)
Description: The five-item Brooding subscale from the Ruminative Responses Scale (RRS) assesses the frequency with which participants experience brooding thoughts in response to depressed mood on a four-point scale from 1 (almost never) to 4 (almost always). An example item is: "People think and do many different things when they feel depressed. Please indicate what you generally do. 'Think what am I doing to deserve this?'" Item scores will be summed to produce an overall score ranging from 5 (min) to 20 (max), where a higher overall score indicates a higher degree of ruminative thoughts (worse outcome).
Time Frame: Measured at baseline and 5 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TGE Individuals
Number analyzed (Participants) | 25
score on a scale
  Baseline | 13.9 (3.60)
  5 months post-baseline: number analyzed (Participants) | 22
  5 months post-baseline | 12.4 (3.24)

ADVERSE EVENTS:
Time Frame: During an assessment or counseling session, from baseline survey to 5-months post-baseline
Arm/Group | TGE Individuals
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 5/25
Other Adverse Events (participants affected / at risk) | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TGE Individuals (N=25)
Suicidal ideation (Psychiatric disorders) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-15): https://cdn.clinicaltrials.gov/large-docs/32/NCT06229132/Prot_SAP_000.pdf